CLINICAL TRIAL: NCT03270033
Title: Analgesic Duration of Interscalene Block After Outpatient Arthroscopic Shoulder Surgery With Intravenous Dexamethasone, Dexmedetomidine or Their Combination: A Randomized Controlled Trial
Brief Title: Intravenous Dexmedetomidine, Dexamethasone and Interscalene Block Duration After Arthroscopic Shoulder Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Manitoba (Other)
Responsible Party: Principal Investigator, Thomas Mutter, Assistant Professor of Anesthesia, University of Manitoba
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B2017:053
Record Dates: First submitted 2017-08-29; First posted 2017-09-01 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Pain, Postoperative; Shoulder Joint Disorder; Ambulatory Surgical Procedures; Brachial Plexus Block
Keywords: Shoulder Joint; Arthroscopy; Ambulatory surgical procedures; Pain, Postoperative; Brachial Plexus Block; Corticosteroid; Dexamethasone; Dexmedetomidine; Bupivacaine; Alpha 2 agonist; Postoperative analgesia
MeSH Terms: conditions — Pain, Postoperative | interventions — Dexamethasone; dexamethasone 21-phosphate; Dexmedetomidine; Injections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dexamethasone (Active Comparator): 4 milligrams dexamethasone administered once intravenously with a 30 millilitres 0.5% bupivacaine interscalene brachial plexus block
  Interventions: Drug: Dexamethasone
- Dexmedetomidine (Active Comparator): 50 micrograms dexmedetomidine administered once intravenously with a 30 millilitres 0.5% bupivacaine interscalene brachial plexus block
  Interventions: Drug: Dexmedetomidine
- Dexamethasone and Dexmedetomidine (Active Comparator): 4 milligrams dexamethasone and 50 micrograms dexmedetomidine administered once intravenously with a 30 millilitres 0.5% bupivacaine interscalene brachial plexus block
  Interventions: Drug: Dexamethasone; Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Dexamethasone — 0.4 millilitres (mL) of 10 milligram per mL sterile, preservative free solution diluted in 50 or 100mL of normal saline and administered once, over approximately 15 minutes, in the immediate preoperative period.
  Other Names: Dexamethasone Omega Unidose (Omega Laboratories Limited); Dexamethasone Sodium Phosphate USP (1 millilitre vial)
  Arms: Dexamethasone; Dexamethasone and Dexmedetomidine
Drug: Dexmedetomidine — 0.5 millilitres (mL) of 100 microgram per mL sterile, preservative free solution diluted in 50 or 100mL of normal saline and administered once, over approximately 15 minutes, in the immediate preoperative period.
  Other Names: Precedex (Hospira Healthcare Corporation); Dexmedetomidine Hydrochloride for Injection
  Arms: Dexamethasone and Dexmedetomidine; Dexmedetomidine

SUMMARY:
In this single-centre, double-blinded, randomized controlled superiority trial, 189 participants having outpatient, arthroscopic shoulder surgery will be randomized into 3 equal sized groups. All participants will receive a standardized interscalene brachial plexus block and 4mg of dexamethasone or 50mcg of dexmedetomidine or both intravenously just prior to their surgery. The purpose of this study is to provide a head to head comparison of two types intravenous adjuncts to ISB, corticosteroids and alpha 2 agonists, and determine if their combination, or either one alone provides superior postoperative analgesia in arthroscopic shoulder surgery patients, as well as possibly show a synergistic relationship between the two adjuncts. The investigators hypothesize the combination of adjuncts will provide a longer duration of analgesia compared to either single agent.

DETAILED DESCRIPTION:
BACKGROUND & RATIONALE Optimal postoperative analgesia is very important in the ambulatory arthroscopic shoulder surgery patient population; interscalene blocks are used for this surgery because they reduce acute pain and have opioid sparing effects postoperatively. While older patients, higher ASA grades and more complex arthroscopic procedures are risk factors for unplanned overnight admissions, in the ambulatory surgery setting, poor analgesia is one of the most common reasons a patient visits a health care provider after their surgery. Approximately 30 % of patients undergoing arthroscopic surgery globally experience significant postoperative pain within the first 24 hours post surgery. In light of this, interscalene brachial plexus blockade (ISB) has been found to be the most effective and preferred method of analgesia for arthroscopic shoulder surgeries when compared to subacromial/intra-articular injections, cryotherapy and oral pain medications. ISB usually consists of a single injection of local anesthetic, anywhere from 5 to 30 minutes prior to shoulder surgery. Although ISB reduces postoperative pain in arthroscopic shoulder surgeries, the length of analgesia from a single injection of local anesthetic is limited to 6 to 15 hours after surgery. Due to the limited duration of analgesia, interscalene catheters have been studied for prolongation of analgesia via continuous infusion of local anesthetics. Although continuous catheter infusions are effective and feasible, there exist several complications such as dyspnea, peripheral neuropathies, nausea, and practical challenges that limit their wider application in an ambulatory setting. Recently, different adjuncts given in combination with local anesthetics have been used to prolong the analgesic duration of a single injection ISB. These adjuncts have been given by both the intravenous and by the perineural routes, where perineural means the adjunct is injected with the local anesthetic around the brachial plexus.

Dexamethasone, a potent glucocorticoid, has been shown in multiple studies to prolong the duration of analgesia of the ISB compared to placebo when administered either perineurally or intravenously. A recently completed large trial (in press) at our centre showed that the duration of analgesia (mean (standard deviation), in hours (h)) with 4mg of intravenous dexamethasone (24.0 (4.6)h) is not significantly different from 8mg (24.8 (6.4)h) and only slightly shorter than perineural dexamethasone doses of 4mg (25.4 (6.6)h) or 8mg (27.2 (8.5)h). The 4mg intravenous dose was favored given the established safety of the intravenous route, its approximately equivalent effectiveness compared to the higher 8mg dose and the absence of differences in adverse effects between groups.

Dexmedetomidine, a highly selective α2 adrenergic agonist with sedative and analgesic properties, has also been shown to potentiate peripheral nerve blockade and prolong the duration of analgesia versus placebo when used as an adjunct to local anesthetic for regional anesthesia, including interscalene block. Most studies have compared perineural dexmedetomidine to placebo, as is the case for other adjuncts such as dexamethasone, even though there is less experience with the perineural route for dexmedetomidine compared to dexamethasone. Interestingly, a recent study found both intravenous and perineural dexmedetomidine reduced the 24 hour opioid consumption and comparably prolonged the duration of ISB analgesia compared to placebo. In a recent meta-analysis, a 50-60ug Dexmedetomidine perineural or intravenous dose maximized sensory block duration while minimizing hemodynamic side effects.

To our knowledge, there are no published studies comparing the analgesic duration of ISB between dexamethasone and dexmedetomidine, and no studies have evaluated whether there is additional benefit to administering these widely available medications in combination. Three ongoing studies are comparing dexamethasone and dexmedetomidine as single adjuncts, without a combination. All three of these studies are using the perineural route, despite the established safety and effectiveness of the intravenous route for both drugs. With this study we are seeking to improve our patients' postoperative experience with superior analgesia by better defining the relative analgesic effectiveness of dexamethasone and dexmedetomidine when given alone or in combination as intravenous adjuncts to ISB.

OBJECTIVES AND HYPOTHESES

In outpatients undergoing arthroscopic shoulder surgery with Interscalene Block:

I. To determine if there is a significant increase in duration of analgesia when combining intravenous dexamethasone and dexmedetomidine compared to administering each adjunct individually. We hypothesize the combination of adjuncts will provide a longer duration of analgesia compared to either single agent.

II. To compare the effect of Dexamethasone to Dexmedetomidine on duration of analgesia when given individually. We hypothesize that there will be no significant difference between the two adjuncts.

METHODS This single-centre, double-blinded, randomized controlled superiority trial has three parallel groups and 1:1:1 randomization. Consenting and eligible adult ambulatory patients undergoing arthroscopic shoulder surgery will receive preoperative, ultrasound guided ISB with 30 millilitres (mL) of 0.5% bupivacaine and 4mg of preservative free dexamethasone or 50mcg of dexmedetomidine or both intravenously. The remainder of the intraoperative and postoperative care is at the discretion of the attending anesthesiologist and surgeon. The primary outcome is analgesic block duration. The power analysis for this study was based on published results from previous studies, as well as our recent work. With a two-tailed alpha error of 0.05, and a standard deviation of 5.0 hours in each group, 180 total patients would provide greater than 90% power to detect a difference of 3.0 hours in block duration. To account for a 5% attrition rate we propose recruiting 63 patients per group (189 patient's total). Outcomes will be assessed by chart review and telephone follow up on postoperative day one, postoperative day 2 (if necessary), and postoperative day 14.

After collecting 102 primary outcomes, we will compare the primary outcome between the combination and each of the single adjuncts. At this point the study will be 90% powered to detect a difference of 6.0h in block duration, even if the standard deviations are higher than expected, at 7.5 hours. If the combination is superior to both of the single agents, the study will be terminated. The principle investigator cancelled this interim analysis on 18 December 2017 after consultation with the study statistician and research team. After reconsidering the original power calculations, the clinically plausible differences between groups, and the high level of statistical significance recommended for interim analyses, it was determined that this interim analysis would be very unlikely to convincingly demonstrate the superiority of the combination over the single agents. As of 18 December 2017 90 patients have participated in the study and recruitment is on schedule. The entire research team has been and will continue to be blinded to outcome data by group assignment until all 189 patients have participated, which is expected to occur in the second quarter of 2018.

The primary outcome analysis will analyze by intention to treat only those patients who were randomized and did receive an attempt at an interscalene block. A secondary analysis will exclude patients who had a "failed" interscalene block in the post anesthesia care unit. A tertiary analysis will be a multivariable analysis adjusted for demographics, preoperative naproxen use, use of general anesthesia, cumulative analgesic use and failed interscalene block.

ELIGIBILITY:
Inclusion Criteria:

* Elective ambulatory surgery patients undergoing arthroscopic shoulder surgery
* Including rotator cuff repair
* Stabilization procedures
* Acromioplasty
* Debridement and distal clavicle excision

Exclusion Criteria:

* Patient refusal
* Diabetes
* Pregnancy
* Coagulopathy significant enough to be a contraindication to regional anesthesia as determined by the attending anesthesiologist
* Sensitivity to local anesthetics, dexamethasone or dexmedetomidine
* Severe chronic obstructive pulmonary disease
* Contralateral vocal cord paralysis
* Contralateral diaphragmatic paralysis
* Surgical limb brachial plexus neuropathy
* Interscalene block site infection
* Systemic glucocorticoids in the last 2 weeks
* Epidural or intraarticular steroid injection in the past 3 months
* Chronic opioid use defined as daily use for the last two weeks
* Active peptic ulcer disease
* End-stage renal disease
* Cirrhotic liver disease
* Ventricular dysfunction
* Advanced heart block
* Previous participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Actual)
Dates: Start 2017-09-18 (Actual); Primary Completion 2018-04-14 (Actual); Study Completion 2018-10-13 (Actual)

PRIMARY OUTCOMES:
Duration of analgesia after ISB | Time-to-event outcome measure, assessed up to the end of postoperative day 3 (approximately 84 hours from performance of the block
  Time from block performance to the first time shoulder pain was experienced after the surgery, rounded to the nearest 0.1 hours, as reported by the participant at telephone follow-up on postoperative day one, or if necessary, postoperative day 2.

SECONDARY OUTCOMES:
Block Success or Failure | Assessed at discharge from the post anesthesia care unit, an expected average of 5 hours after the performance of the block.
  The block will be considered "failed" if the patient required opioid analgesia for surgical site pain during their stay in the post anesthesia care unit, as determined by the patient's nurse. At our facility, patients are discharged home directly from the post anesthesia care unit.
Cumulative Analgesic Consumption in the post anesthesia care unit | "Change" outcome measure: From admission to the post anesthesia care unit (an expected average of 2.5 hours after performance of the block), to discharge from the post anesthesia care unit (an expected average of 4 hours after performance of the block)
  Measured as equivalent milligrams of morphine
Cumulative Analgesic Consumption from post anesthesia care unit discharge until the time the primary outcome occurred | "Change" outcome measure: From discharge from the post anesthesia care unit (an expected average of 5 hours after performance of the block), to the occurrence of the primary outcome (an expected average of 28 hours after performance of the block)
  Measured as equivalent milligrams of morphine
Unplanned Postoperative Hospital Admission, as reported at telephone follow up or chart review | Assessed at telephone follow up on postoperative day one and chart review
  Transfer or admission to hospital during the postoperative period between admission to the post anesthesia care unit and telephone follow up on postoperative day one
New Persistent Neurologic Symptoms | Assessed at postoperative day 14
  Patient will be asked whether they are experiencing any tingling, numbness or weakness in the surgical limb, or hoarseness or dyspnea. Patients answering yes to any of the above will have a detailed telephone assessment and be reassessed by telephone at 6 months postoperatively
Post anesthesia care unit length of stay in minutes | Assessed at discharge from the post anesthesia care unit, an expected average of 4 hours after performance of the block.
  Amount of time between admission and discharge from the post anesthesia care unit.
The QoR-15 questionnaire | Assessed at postoperative day one.
  A standardized and validated 15 item questionnaire consisting exclusively of 11 point integer scale questions (10 = all the time, 0 = none of the time) designed to assess quality of recovery, physical and mental wellbeing in patients recovering from surgery. A total composite score is measured as the total of all 15 individual scores.

OTHER OUTCOMES:
Intraoperative and post anesthesia care unit use of cardiovascular medications, as recorded in the patient's chart | Assessed at discharge from the post anesthesia care unit, an expected average of 4 hours after the performance of the block
  The use of Intraoperative vasopressors, inotropes, antimuscarinics or antihypertensives at any time between the performance of the block and discharge from the post anesthesia care unit
Adverse events previously related to the inter scalene block and unlikely related to dexamethasone or dexmedetomidine, as recorded in the patient's chart. | Assessed at discharge from the post anesthesia care unit, an expected average of 4 hours after the performance of the block
  The occurrence of seizure, systemic local anesthetic toxicity, pneumothorax, hemothorax, epidural spread of local anesthetic, or hoarse voice at any time between the performance of the block and discharge from the post anesthesia care unit.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas C Mutter, MD MSc, Principal Investigator — Assistant Professor
Locations (1):
- Pan Am Surgical Centre, Winnipeg, Manitoba, Canada

REFERENCES:
- [Background] Brattwall M, Jildenstal P, Warren Stomberg M, Jakobsson JG. Upper extremity nerve block: how can benefit, duration, and safety be improved? An update. F1000Res. 2016 May 18;5:F1000 Faculty Rev-907. doi: 10.12688/f1000research.7292.1. eCollection 2016. PMID 27239291
- [Background] Sultan J, Marflow KZ, Roy B. Unplanned overnight admissions in day-case arthroscopic shoulder surgery. Surgeon. 2012 Feb;10(1):16-9. doi: 10.1016/j.surge.2010.11.033. Epub 2011 Jan 20. PMID 22233552
- [Background] Fortier J, Chung F, Su J. Unanticipated admission after ambulatory surgery--a prospective study. Can J Anaesth. 1998 Jul;45(7):612-9. doi: 10.1007/BF03012088. PMID 9717590
- [Background] Hughes MS, Matava MJ, Wright RW, Brophy RH, Smith MV. Interscalene brachial plexus block for arthroscopic shoulder surgery: a systematic review. J Bone Joint Surg Am. 2013 Jul 17;95(14):1318-24. doi: 10.2106/JBJS.L.01116. No abstract available. PMID 23864181
- [Background] Warrender WJ, Syed UAM, Hammoud S, Emper W, Ciccotti MG, Abboud JA, Freedman KB. Pain Management After Outpatient Shoulder Arthroscopy: A Systematic Review of Randomized Controlled Trials. Am J Sports Med. 2017 Jun;45(7):1676-1686. doi: 10.1177/0363546516667906. Epub 2016 Oct 13. PMID 27729319
- [Background] Fredrickson MJ, Krishnan S, Chen CY. Postoperative analgesia for shoulder surgery: a critical appraisal and review of current techniques. Anaesthesia. 2010 Jun;65(6):608-624. doi: 10.1111/j.1365-2044.2009.06231.x. PMID 20565394
- [Background] Fredrickson MJ, Leightley P, Wong A, Chaddock M, Abeysekera A, Frampton C. An analysis of 1505 consecutive patients receiving continuous interscalene analgesia at home: a multicentre prospective safety study. Anaesthesia. 2016 Apr;71(4):373-9. doi: 10.1111/anae.13385. Epub 2016 Feb 5. PMID 26849172
- [Background] Marhofer P, Anderl W, Heuberer P, Fritz M, Kimberger O, Marhofer D, Klug W, Blasl J. A retrospective analysis of 509 consecutive interscalene catheter insertions for ambulatory surgery. Anaesthesia. 2015 Jan;70(1):41-6. doi: 10.1111/anae.12840. Epub 2014 Sep 10. PMID 25209310
- [Background] YaDeau JT, Gordon MA, Goytizolo EA, Lin Y, Fields KG, Goon AK, Holck G, Miu TW, Gulotta LV, Dines DM, Craig EV. Buprenorphine, Clonidine, Dexamethasone, and Ropivacaine for Interscalene Nerve Blockade: A Prospective, Randomized, Blinded, Ropivacaine Dose-Response Study. Pain Med. 2016 May;17(5):940-60. doi: 10.1093/pm/pnv010. Epub 2015 Dec 14. PMID 26814246
- [Background] Chalifoux F, Colin F, St-Pierre P, Godin N, Brulotte V. Low dose intravenous dexamethasone (4 mg and 10 mg) significantly prolongs the analgesic duration of single-shot interscalene block after arthroscopic shoulder surgery: a prospective randomized placebo-controlled study. Can J Anaesth. 2017 Mar;64(3):280-289. doi: 10.1007/s12630-016-0796-6. Epub 2017 Jan 3. PMID 28050801
- [Background] Routman HD, Israel LR, Moor MA, Boltuch AD. Local injection of liposomal bupivacaine combined with intravenous dexamethasone reduces postoperative pain and hospital stay after shoulder arthroplasty. J Shoulder Elbow Surg. 2017 Apr;26(4):641-647. doi: 10.1016/j.jse.2016.09.033. Epub 2016 Nov 15. PMID 27856266
- [Background] Webb BG, Sallay PI, McMurray SD, Misamore GW. Comparison of Interscalene Brachial Plexus Block Performed With and Without Steroids. Orthopedics. 2016 Nov 1;39(6):e1100-e1103. doi: 10.3928/01477447-20160819-02. Epub 2016 Aug 30. PMID 27575034
- [Background] Rosenfeld DM, Ivancic MG, Hattrup SJ, Renfree KJ, Watkins AR, Hentz JG, Gorlin AW, Spiro JA, Trentman TL. Perineural versus intravenous dexamethasone as adjuncts to local anaesthetic brachial plexus block for shoulder surgery. Anaesthesia. 2016 Apr;71(4):380-8. doi: 10.1111/anae.13409. Epub 2016 Feb 22. PMID 26899862
- [Background] Desmet M, Vanneste B, Reynvoet M, Van Cauwelaert J, Verhelst L, Pottel H, Missant C, Van de Velde M. A randomised controlled trial of intravenous dexamethasone combined with interscalene brachial plexus blockade for shoulder surgery. Anaesthesia. 2015 Oct;70(10):1180-5. doi: 10.1111/anae.13156. Epub 2015 Jun 17. PMID 26082203
- [Background] Jadon A, Dixit S, Kedia SK, Chakraborty S, Agrawal A, Sinha N. Interscalene brachial plexus block for shoulder arthroscopic surgery: Prospective randomised controlled study of effects of 0.5% ropivacaine and 0.5% ropivacaine with dexamethasone. Indian J Anaesth. 2015 Mar;59(3):171-6. doi: 10.4103/0019-5049.153039. PMID 25838589
- [Background] Woo JH, Kim YJ, Kim DY, Cho S. Dose-dependency of dexamethasone on the analgesic effect of interscalene block for arthroscopic shoulder surgery using ropivacaine 0.5%: A randomised controlled trial. Eur J Anaesthesiol. 2015 Sep;32(9):650-5. doi: 10.1097/EJA.0000000000000213. PMID 25603389
- [Background] Fritsch G, Danninger T, Allerberger K, Tsodikov A, Felder TK, Kapeller M, Gerner P, Brummett CM. Dexmedetomidine added to ropivacaine extends the duration of interscalene brachial plexus blocks for elective shoulder surgery when compared with ropivacaine alone: a single-center, prospective, triple-blind, randomized controlled trial. Reg Anesth Pain Med. 2014 Jan-Feb;39(1):37-47. doi: 10.1097/AAP.0000000000000033. PMID 24317234
- [Background] Bengisun ZK, Ekmekci P, Akan B, Koroglu A, Tuzuner F. The effect of adding dexmedetomidine to levobupivacaine for interscalene block for postoperative pain management after arthroscopic shoulder surgery. Clin J Pain. 2014 Dec;30(12):1057-61. doi: 10.1097/AJP.0000000000000065. PMID 24366001
- [Background] Abdallah FW, Dwyer T, Chan VW, Niazi AU, Ogilvie-Harris DJ, Oldfield S, Patel R, Oh J, Brull R. IV and Perineural Dexmedetomidine Similarly Prolong the Duration of Analgesia after Interscalene Brachial Plexus Block: A Randomized, Three-arm, Triple-masked, Placebo-controlled Trial. Anesthesiology. 2016 Mar;124(3):683-95. doi: 10.1097/ALN.0000000000000983. PMID 26649424
- [Background] Velazquez-Delgado E, Gaspar-Carrillo SP, Pena-Riveron AA, Mejia-Terrazas GE. Postoperative analgesia with dexmedetomidine in interscalene block. Comparative study. Rev Esp Anestesiol Reanim. 2017 Mar;64(3):137-143. doi: 10.1016/j.redar.2016.07.005. Epub 2016 Sep 9. English, Spanish. PMID 27616331
- [Background] Vorobeichik L, Brull R, Abdallah FW. Evidence basis for using perineural dexmedetomidine to enhance the quality of brachial plexus nerve blocks: a systematic review and meta-analysis of randomized controlled trials. Br J Anaesth. 2017 Feb;118(2):167-181. doi: 10.1093/bja/aew411. PMID 28100520
- [Background] Keplinger M, Marhofer P, Kettner SC, Marhofer D, Kimberger O, Zeitlinger M. A pharmacodynamic evaluation of dexmedetomidine as an additive drug to ropivacaine for peripheral nerve blockade: A randomised, triple-blind, controlled study in volunteers. Eur J Anaesthesiol. 2015 Nov;32(11):790-6. doi: 10.1097/EJA.0000000000000246. PMID 25695189
- [Background] Schulz KF, Altman DG, Moher D. CONSORT 2010 statement: Updated guidelines for reporting parallel group randomised trials. J Pharmacol Pharmacother. 2010 Jul;1(2):100-7. doi: 10.4103/0976-500X.72352. No abstract available. PMID 21350618
- [Background] Montefiore Medical Center; Bronx, New York. The Analgesic Duration of Dexmedetomidine Compared to Dexamethasone as Adjuncts to Single Shot Interscalene Block In: ClinicalTrials.gov [Internet]. Bethesda (MD): National Library of Medicine (US). 2016- [cited 2017 March 5]. Available from: https://clinicaltrials.gov/ct2/show/NCT02653144 NLM Identifier: NCT02653144
- [Background] B. P. Koirala Institute of Health Sciences; Dharan, Sunsari, Nepal. Dexamethasone Compared With Dexmedetomidine as an Adjuvant to Ropivacaine for Supraclavicular Brachial Plexus Block In: ClinicalTrials.gov [Internet]. Bethesda (MD): National Library of Medicine (US). 2016- [cited 2017 March 5]. Available from: https://clinicaltrials.gov/ct2/show/NCT02787018 NLM Identifier: NCT02787018
- [Background] Government Medical College and Hospital; Department of Anaesthesia and Intensive Care, Government Medical and Hospital, Chandigarh, India. A randomised double blind study comparing dexmedetomidine with dexamethasone as an adjunct to ropivacaine in ultrasound guided interscalene block for shoulder surgery In: Clinical Trials Registry India [Internet]. New Delhi: database publisher (India). 2015- [cited 2017 March 5]. Available from: http://www.ctri.nic.in/Clinicaltrials/pmaindet2.php?trialid=11447 Identifier: CTRI/2015/08/006124
- [Background] Waldron NH, Jones CA, Gan TJ, Allen TK, Habib AS. Impact of perioperative dexamethasone on postoperative analgesia and side-effects: systematic review and meta-analysis. Br J Anaesth. 2013 Feb;110(2):191-200. doi: 10.1093/bja/aes431. Epub 2012 Dec 5. PMID 23220857
- [Background] Stark PA, Myles PS, Burke JA. Development and psychometric evaluation of a postoperative quality of recovery score: the QoR-15. Anesthesiology. 2013 Jun;118(6):1332-40. doi: 10.1097/ALN.0b013e318289b84b. PMID 23411725
- [Derived] Rodrigues D, Amadeo RJJ, Wolfe S, Girling L, Funk F, Fidler K, Brown H, Leiter J, Old J, MacDonald P, Dufault B, Mutter TC. Analgesic duration of interscalene block after outpatient arthroscopic shoulder surgery with intravenous dexamethasone, intravenous dexmedetomidine, or their combination: a randomized-controlled trial. Can J Anaesth. 2021 Jun;68(6):835-845. doi: 10.1007/s12630-021-01942-2. Epub 2021 Feb 18. PMID 33598889